CLINICAL TRIAL: NCT03445949
Title: Optimal Antiplatelet Treatment to Achieve Stroke Avoidance and Fall in Bleeding Events Following Left Atrial Appendage Closure (SAFE-LAAC). Comparative Health Effectiveness Randomized Trial - PILOT Study
Brief Title: Optimal Antiplatelet Therapy Following Left Atrial Appendage Closure
Acronym: SAFE-LAAC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.52/IV/16
Record Dates: First submitted 2018-02-01; First posted 2018-02-26 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation, stroke, bleeding, left atrial appendage
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — Long-Term Care; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30 days DAPT and long-term treatment with a single antiplatelet agent (Other): short postimplantation dual antiplatelet therapy and long-term treatment with a single antiplatelet agent
  Interventions: Drug: short postimplantation dual antiplatelet therapy; Drug: long-term treatment with a single antiplatelet agent
- 6 months DAPT and long-term treatment with a single antiplatelet agent (Other): extended postimplantation dual antiplatelet therapy and long-term treatment with a single antiplatelet agent
  Interventions: Drug: extended postimplantation dual antiplatelet therapy; Drug: long-term treatment with a single antiplatelet agent
- 30 days DAPT and 6 months treatment with a single antiplatelet agent (Other): short postimplantation dual antiplatelet therapy and 6 months treatment with a single antiplatelet agent
  Interventions: Drug: short postimplantation dual antiplatelet therapy; Drug: 6 months treatment with a single antiplatelet agent
- 6 months DAPT and 6 months treatment with a single antiplatelet agent (Other): extended postimplantation dual antiplatelet therapy and 6 months treatment with a single antiplatelet agent
  Interventions: Drug: extended postimplantation dual antiplatelet therapy; Drug: 6 months treatment with a single antiplatelet agent

INTERVENTIONS:
Drug: short postimplantation dual antiplatelet therapy — continuing dual antiplatelet therapy up until 6 months after left atrial appendage occlusion with Amplatzer or WATCHMAN device
  Arms: 30 days DAPT and 6 months treatment with a single antiplatelet agent; 30 days DAPT and long-term treatment with a single antiplatelet agent
Drug: extended postimplantation dual antiplatelet therapy — stopping dual antiplatelet therapy after 30 days after left atrial appendage occlusion with Amplatzer or WATCHMAN device
  Arms: 6 months DAPT and 6 months treatment with a single antiplatelet agent; 6 months DAPT and long-term treatment with a single antiplatelet agent
Drug: long-term treatment with a single antiplatelet agent — continuing long-term treatment with single antiplatelet agent
  Arms: 30 days DAPT and long-term treatment with a single antiplatelet agent; 6 months DAPT and long-term treatment with a single antiplatelet agent
Drug: 6 months treatment with a single antiplatelet agent — continuing single antiplatelet agent up until 6 months
  Arms: 30 days DAPT and 6 months treatment with a single antiplatelet agent; 6 months DAPT and 6 months treatment with a single antiplatelet agent

SUMMARY:
SAFE-LAAC Trial has been designed to gather data on the most optimal strategy of antiplatelet therapy after transcatheter left atrial appendage occlusion with Amplatzer or WATCHMAN device

DETAILED DESCRIPTION:
Background:

Transcatheter left atrial appendage closure (LAAC) has been shown to be non-inferior to oral anticoagulation in preventing cardioembolic strokes associated with atrial fibrillation. However, an optimal antithrombotic treatment regimen following successful LAAC remains an unresolved issue. The scope and duration of antiplatelet treatment following LAAC are of paramount importance as they may significantly contribute to post-procedural as well as long-term procedural safety and efficacy.

Objective:

SAFE-LAAC Trial has been designed as a comparative health effectiveness study with the following aims:

1. compare the safety and efficacy of 30 days vs. 6 months of dual antiplatelet therapy following LAAC with Amplatzer or WATCHMAN device (randomized comparison)
2. compare safety and efficacy of stopping all antithrombotic and antiplatelet agents 6 months after LAAC vs. long-term treatment with a single antiplatelet agent (nonrandomized comparison)

Patient population:

Patients (n=200) after successful LAAC with Amplatzer or WATCHMAN device.

Perspective:

Results of this pilot trial will provide: 1. data to aid practitioners and guideline writers recommend the most optimal antithrombotic treatment after LAAC, and 2. data to support power calculations for designing future randomized trials.

Methodology:

SAFE LAAC has been designed as a multicenter (planned contribution of 7 centers in Poland), open-label, comparative health effectiveness trial with central, independent adjudication of events comprising the primary end-point. The first part of the trial is randomized and after 6 months of follow-up continues for another 12 months as a non-randomized study.

Timeline:

The duration of the trial has been planned for 5 years. The enrollment phase has been planned for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Successful left atrial appendage occlusion with Amplatzer or WATCHMAN device within 37 days before randomization
* Treatment with dual antiplatelet therapy (clopidogrel and acetylsalicylic acid) between left atrial appendage closure and randomization
* Participant's age 18 years or older at the time of signing the informed consent form
* Participant is willing to follow all study procedures; especially the randomized antiplatelet treatment regimen
* Participant is willing to sign the study informed consent form

Exclusion Criteria:

* Indications to dual antiplatelet therapy other than atrial fibrillation and/or left atrial appendage occlusion at the time of enrollment or predicted appearance of such indications within the duration of the trial (e.g. planned coronary revascularization)
* Indications to anticoagulation at the time of enrollment and/or predicted appearance of such indications within the duration of the trial (e.g. pulmonary embolism)
* Known allergy to clopidogrel and/or acetylsalicylic acid precluding its administration as specified by the protocol
* Any known inborn or acquired coagulation disorders
* Peridevice leak >5mm on imaging study preceding enrollment
* Left atrial thrombus on an imaging study performed after successful left atrial appendage closure but before enrollment
* Life expectancy of fewer than 18 months
* Participation in other clinical studies with experimental therapies at the time of enrollment and preceding 3 months
* Chronic kidney disease stage IV and V
* Women who are pregnant or breastfeeding; women of childbearing potential who do not consent to apply at least two methods of contraception. This criterion does not apply to women 2 years post menopause (with negative pregnancy test 24 hours prior to randomization if <55 years old) or after surgical sterilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2025-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Efficacy (a composite of ischemic stroke, transient ischaemic attack, peripheral embolism, nonfatal myocardial infarction, cardiovascular mortality, all-cause mortality, left atrial appendage thrombus) | 17 months
  Event rates reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Safety (moderate and/or severe bleeding (BARC type 2, 3, and 5) | 17 months
  Event rates reported per 100 patient-years (calculated as 100*N events/Total patient-years);

SECONDARY OUTCOMES:
Ischemic stroke | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Transient ischaemic attack | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Peripheral embolism | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Nonfatal myocardial infarction | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Cardiovascular mortality | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
All-cause mortality | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Moderate and/or severe bleeding (BARC type 2,3, and 5) | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Left atrial appendage thrombus | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
Any bleeding | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years);
New moderate or major (≥4 mm) ischemic brain lesions on magnetic resonance imaging | 17 months
  Event rate reported per 100 patient-years (calculated as 100*N events/Total patient-years)
Change in cognition score as detected by the Addenbrooke's cognitive examination (ACE-III) | 17 months
  ACE-III is a screening test that is composed of tests of attention, orientation, memory, language, visual perceptual, and visuospatial skills. The total range of raw score is 0-100. A higher score indicates more intact cognitive functioning

OTHER OUTCOMES:
Number of new ischemic brain lesions on magnetic resonance imaging | 17 months
Volume of new ischemic brain lesions on magnetic resonance imaging | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Pracon, MD PhD, Principal Investigator — Coronary and Structural Heart Diseases Department, National Institute of Cardiology, Warsaw, Poland; Marcin Demkow, MD PhD, Principal Investigator — Coronary and Structural Heart Diseases Department, National Institute of Cardiology, Warsaw, Poland
Locations (1):
- National Institute of Cardiology, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided